CLINICAL TRIAL: NCT07402512
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of Deurremidevir Hydrobromide for Oral Suspension in Infants and Young Children With Respiratory Syncytial Virus Infection
Brief Title: A Phase III Clinical Trial on the Efficacy and Safety of Deuremidevir Hydrobromide Dry Suspension for the Treatment of RSV Infection in Infants and Young Children
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0916-301
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIM0916 (Experimental)
  Interventions: Drug: SIM0916
- SIM0916 Placebo (Placebo Comparator)
  Interventions: Drug: SIM0916 Placebo

INTERVENTIONS:
Drug: SIM0916 — Dose: 20 mg/kg TID
  Arms: SIM0916
Drug: SIM0916 Placebo — Dose: 20 mg/kg TID
  Arms: SIM0916 Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group trial conducted in infants and young children aged 1 to 36 months with RSV infection.

A total of 498 subjects are expected to be enrolled and randomly assigned to the investigational product group or the placebo group in a 2:1 ratio; Administration will be based on the subject's weight, with a dose of 20 mg/kg three times daily for 5 consecutive days (15 doses).

ELIGIBILITY:
Inclusion Criteria:

1. Infants and young children aged ≥ 1 month and ≤ 36 months, regardless of gender;
2. Weight ≥ 2.5 kg and ≤ 20 kg;
3. Positive RSV antigen or nucleic acid test
4. Duration of illness due to RSV infection ≤ 96 hours;
5. Presence of tachypnea and wheezing;
6. Wang Bronchiolitis Score≥ 5;
7. For subjects aged < 12 months, head circumference should be within the normal range corresponding to their age and gender.

Exclusion Criteria:

1. Subjects who have received protocol-speciﬁed prohibited medications:
2. Subjects with severe intrapulmonary complications or extrapulmonary complications;
3. Subjects requiring vasopressors or inotropic agents;
4. Subjects with known concurrent SARS-CoV-2 infection, inﬂuenza virus infection, Mycoplasma infection, or suspected concurrent bacterial or other pathogen infections;
5. Subjects with a known history of hypercapnia;
6. Subjects with chronic or persistent feeding diﬃculties;
7. Subjects with gastrointestinal diseases that the investigator believes may signiﬁcantly aﬀect the absorption of the study drug;
8. Subjects with congenital metabolic abnormalities;
9. Subjects with bronchopulmonary dysplasia requiring assisted ventilation or clinically signiﬁcant congenital respiratory tract abnormalities;
10. Subjects with congenital heart disease (CHD) that the investigator assesses may aﬀect eﬃcacy evaluation;
11. Subjects with clinical evidence of hepatic decompensation; or abnormal liver function tests;
12. Subjects with renal failure, including renal abnormalities potentially related to renal insuﬃciency or abnormal renal function tests;
13. Subjects with a known history of HIV positivity, or suspected to be HIV positive by the investigator;
14. Subjects with known or suspected primary immunodeﬁciency diseases or transplant recipients;
15. Subjects with a history of epilepsy or febrile convulsions;
16. Subjects with a personal or family history of severe allergies or allergies;
17. Subjects with active or uncontrolled respiratory, cardiac, hepatic, central nervous system, or renal diseases, or other medical conditions deemed unsuitable for enrollment by the investigator;
18. Subjects who participated in other drug or medical device clinical trials and received investigational products or devices;
19. Subjects deemed unsuitable for participation in this study by the investigator for any other reason.

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 498 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The earliest time from the first dose to the sustained resolution of 6 RSV infection-related clinical signs and symptoms | Day 26
  The earliest time from the first dose to the sustained resolution of 6 RSV infection-related clinical signs and symptoms. Resolution of 6 RSV infection-related clinical signs and symptoms is defined as a score of 0 for all of 6 RSV infection-related clinical signs.

SECONDARY OUTCOMES:
The earliest time from the first dose to the sustained relief/resolution of wheezing.Relief/resolution of wheezing is defined as a wheezing score ≤ 1. | Day 26
Change in Wang Bronchiolitis Score from baseline on Days 2-6 and Day 14 after the first dose | Day 26
Time from the first dose to disease recovery: the earliest time when Wang Bronchiolitis Score ≤ 1 | Day 26
Proportion of subjects achieving RSV disease recovery (Wang Bronchiolitis Score ≤ 1 at daily assessment) on each day from Day 2 to Day 6 and on Day 14 after the first dose | Day 26
Earliest time from the first dose to the sustained resolution of individual RSV infection-related clinical signs and symptoms | Day 26
Proportion of subjects with resolution of individual RSV infection-related clinical signs and symptoms | Day 26
Proportion of subjects with wheezing score ≤ 1 at daily assessment on each day from Day 2 to Day 6 and on Day 14 after the first dose; | Day 26
Time from the first dose to the sustained relief/resolution of cough. Relief/resolution of cough is defined as a cough score ≤ 1 | Day 26
Proportion of subjects with cough score ≤ 1 at daily assessment on each day from Day 2 to Day 6 and on Day 14 after the first dose | Day 26
Number and duration of admissions to the Intensive Care Unit (ICU) due to RSV infection-related diseases; | Day 26
Number of times of non-invasive positive pressure ventilation or mechanical ventilation received due to RSV infection-related diseases | Day 26

OTHER OUTCOMES:
Change in viral load from baseline on Days 2-6 and Day 14 after the first dose | Day 26
Proportion of subjects with viral load below the Lower Limit of Quantitation (LLOQ) on Days 2-6 and Day 14 after the first dose | Day 26
Area under the viral load-time curve from baseline to Days 2-6 and Day 14 after the first dose | Day 26

CONTACTS AND LOCATIONS:
Overall Officials: hanmin liu, Principal Investigator — West China Second University Hospital; lanjuan Li, Principal Investigator — Shulan (Hangzhou) Hospital
Locations (2):
- China (2):
  - West China Second University Hospital Sichuan University, Chengdu, Sichuan
  - Shulan(hangzhou)Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No